## Seating System for Scoliosis in Non-ambulatory Children with Cerebral Palsy:

## **A Randomized Controlled Trial**

Clinical trials number: NCT03862625

Date of Data: 02.02.2019

## **Statistical Analysis Plan**

Statistical analysis was performed using the IBM SPSS version 23.0 software (Statistics for MacOs, IBM Corp., Armonk, NY, USA). This is a pilot study since no similar studies have been identified. Descriptive statistics of data were expressed in mean and standard deviation values in parametric tests; median, minimum and maximum values in non parametric tests. The Shapiro-Wilk test was used to analyze whether the data were normally distributed. The Wilcoxon paired-samples test was used to analyze the data which were not normally distributed. In comparison of BT and AT values, Wilcoxon Signed Ranks test was used for paired measurements. The difference between the values obtained before and after the treatment (posttest-pretest) was calculated and Mann Whitney U test was used to compare this difference between the groups. For the sample size, the confidence interval was %95 and p value of < 0,05 was considered statistically significant.